CLINICAL TRIAL: NCT06215573
Title: Effect of a Novel Melatonin Supplement on Sleep Quality
Acronym: I-MASQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Ritual Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: WT4634027_I-MASQ v2.0
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sleep
Keywords: melatonin; pharmacokinetics; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomised cross over trial counterbalanced for trial order
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Coded, known only to manufacturer / collaborator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin supplementation (Experimental): 5mg melatonin supplement from Ritual Inc's BioSeries
  Interventions: Dietary Supplement: Melatonin
- Placebo supplementation (Placebo Comparator): Placebo supplement from Ritual Inc.
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Melatonin — 5mg melatonin supplement, once daily, from Ritual BioSeries
  Arms: Melatonin supplementation
Dietary Supplement: Placebo supplement — Placebo supplement, once daily, from Ritual BioSeries
  Arms: Placebo supplementation

SUMMARY:
Melatonin is a hormone naturally found in our body that increases in our blood at night and controls how we sleep. Melatonin can also be taken as a pill and numerous clinical trials have documented improved sleep quality following melatonin supplementation before bed. However, it is not known whether such supplements actually increase blood melatonin above normal levels, particularly at night.

The aims of this study are to investigate whether a novel melatonin supplement (Ritual Sleep BioSeriesTM Melatonin) can increase blood melatonin in human participants at night, and to determine if taking the supplement before bed for two-weeks can improve sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Aged 18-40
* Sometimes have trouble sleeping (Pittsburgh sleep quality index score >5)

Exclusion Criteria:

* Routinely taking melatonin supplements or other drugs known to affect sleep
* A diagnosed sleep disorder
* Major psychiatric illness
* Current physical injury
* Known or suspected hypersensitivity to melatonin
* Presence of major sleep disruptors at home (e.g. new born baby)
* Night shift/rotational-shift work
* Receiving non-pharmacological treatment for sleep disorder (e.g. cognitive behavioral therapy)
* Substance use disorder
* Recent (<1 month) increase in daily caffeinated drink consumption
* Consuming >14 standard alcoholic drinks per week
* Pregnant or lactating

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic | 10 hours
  Serum melatonin concentration area under curve
Sleep efficiency | 2 weeks
  Sleep efficiency, as total time asleep as percentage of time in bed

SECONDARY OUTCOMES:
Sleep diary | 2 weeks
  Sleep diary recorded daily via 'consensus sleep diary - core'
Recovery and well being | 2 weeks
  Recovery and well being recorded via recovery stress questionnaire (REST-Q)
Sleep quality | 2 weeks
  Sleep quality determined via 'Pittsburgh Sleep Quality Index survey'

CONTACTS AND LOCATIONS:
Overall Officials: Francis B Stephens, PhD, Principal Investigator — University of Exeter
Locations (1):
- Sport & Health Sciences University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No